CLINICAL TRIAL: NCT02539082
Title: A Post-marketing Surveillance to Evaluate the Safety and Efficacy of Collagen Injection in Patients With Plantar Fasciitis
Brief Title: the Safety and Efficacy of Collagen Injection in Patients With Plantar Fasciitis
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sewon Cellontech Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 01RGS
Record Dates: First submitted 2015-08-31; First posted 2015-09-02 (Estimated); Last update posted 2015-09-02 (Estimated); Status verified 2015-08

CONDITIONS: Plantar Fasciitis
Keywords: collagen; collagen injection; plantar fasciitis
MeSH Terms: conditions — Fasciitis, Plantar | interventions — Saline Solution

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- placebo injection (Placebo Comparator): placebo, normal saline, injection in the plantar facia through randomization
  Interventions: Drug: normal saline
- Regenseal injection (Experimental): Regenseal, collagen, injection in the plantar facia through randomization
  Interventions: Device: Regenseal

INTERVENTIONS:
Device: Regenseal — Regenseal, collagen, injection in the defect area
  Arms: Regenseal injection
Drug: normal saline — placebo, normal saline, injection in the defect area
  Arms: placebo injection

SUMMARY:
The primary objective of this study is to evaluate the safety and efficacy of collagen injection in patients with plantar fasciitis

DETAILED DESCRIPTION:
This study is an open-trial study. Sixty subjects will be participated in it. The study will be explained to the subjects and they voluntarily agreed to participate in it. Their eligibility to participate in the study will be checked, and the patient will receive collagen or a placebo (normal saline) in the plantar facia through randomization. They will be asked to follow the guidelines of the investigators during the study and to visit the hospital seven times, including for screening and the date of re-injection. . At each visit, the subjects undergo a VAS, a clinical laboratory tests, and a physical exam to evaluate the safety and efficacy of Regenseal. (*Re-injection could be maximum 2times at visit2 and 3, one week apart based on the investigator's judgment after the initial injection. If the subject gets injection on the screening date, the total number of his or her visits will be six.)

ELIGIBILITY:
Inclusion Criteria:

- 1. Patient with chronic plantar fasciitis (Patients who had been diagnosed with plantar fasciitis but had not been responsive to non-invasive treatment for more than three months (non-invasive treatments include drugs, physiotherapy shock wave, or stretching) 2. Patients who are able to complete the questionnaires related to the safety and efficacy of the study drug and who read and understood the guidelines 3. Patients who agreed to maintain the medication dose during the study period if they need to keep taking it. (Excluded anti-inflammatory analgesic drug for pain after the injection.) 4. Patients who agreed not to use physical therapy or shock wave during the study period.

5. Patients or their representative (for adults), or patients and their parent/guardian (for minors), who agreed to participate in the study and signed the informed consent form

Exclusion Criteria:

* 1. If patients or their families suffer from or have ever suffered from an autoimmune disease.

  2. Patients who have ever suffered an anaphylactic reaction. 3. Patients who have ever suffered hypersensitivity to an implant. 4. Patients with a history of allergy to porcine or bovine protein. 5. Patients with rheumatoid arthritis. 6. Patients with ankylosing spondylitis. 7. Patients who are suspected of having spinal deformity with a negative serum test 8. Subjects who are pregnant and/or breast-feeding and/or plan a pregnancy. 9. Subjects with psychiatric disorders who are considered inappropriate to participate in this trial by the Principal Investigator.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2013-11; Primary Completion 2016-04 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
The difference in the 100mmVAS score | 3 months after the surgery
  The difference in the 100mmVAS between study group and control group at 3 months after the surgery will be compared and analyzed

SECONDARY OUTCOMES:
The difference in the 100mmVAS score | baseline and 6, 12 months after the surgery
  The difference in the 100mmVAS between study group and control group at baseline and 6, 12 months after the surgery will be compared and analyzed.
change of the thickness in the sonographic evaluation and fluid collection | baseline and 3, 6, 12 months after the surgery
  The difference between study group and control group of the thickness in the sonographic evaluation and fluid collection at baseline will be compared with that three months after the surgery. The thickness in the sonographic evaluation and fluid collection six and 12 months will be additionally taken for comparison and analysis.
change of Satisfaction evaluation by physician in charge | baseline and 3, 6, 12 months after the surgery
  The improvements on the affected ankle by physician in charge at 3 months after injection and six, 12months after injection of the study and control group will be compared and analyzed. (Physician in charge evaluates the degree of improvement in 5 levels, such as 'excellent, good, satisfactory, no change, and worsened.)
change of Satisfaction evaluation by patients | baseline and 3, 6, 12 months after the surgery
  The improvements on the affected ankle at 3 months after injection and six, 12 months after injection of the study and control group will be compared and analyzed. (Patient evaluates the degree of improvement in 5 levels, such as 'excellent, good, satisfactory, no change, and worsened.)
change score of Degree of recovery | baseline and 3, 6, 12 months after the surgery
  The score of degree of recovery at baseline will be recorded. The difference between study group and control group in the score of degree of recovery at three, six, and 12months after injection will be compared and analyzed.

CONTACTS AND LOCATIONS:
Overall Officials: Jin Soo Kim, MD, Principal Investigator — Eulji General Hospital; Jae Ho Cho, MD, Principal Investigator — Inje University; Jun Bum Kim, MD, Principal Investigator — Daejeon Sun Hospital
Locations (3):
- South Korea (3):
  - Daejeon Sun Hospital, Daejeon, Daejeon
  - Eulji General Hospital, Seoul, Seoul
  - Inje University Seoul Paik Hospital, Seoul, Seoul